CLINICAL TRIAL: NCT00346320
Title: A Phase II Study of Accelerated Hypofractionated 3-Dimensional Conformal Radiotherapy (3DCRT) For Inoperable Stage I/II Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Radiation in Stage I or Stage II Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR25; CAN-NCIC-BR25 (Other: PDQ); CDR0000486919 (Other: PDQ)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): 3-dimensional conformal radiotherapy, 60 Gy in once daily 4 Gy fractions (Monday to Friday) over 3 weeks
  Interventions: Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — 3-dimensional conformal radiotherapy, 60 Gy in once daily 4 Gy fractions (Monday to Friday) over 3 weeks

SUMMARY:
RATIONALE: Radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well radiation therapy works in treating patients with stage I or stage II non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the local tumor control rate at 2 years after accelerated hypofractionated 3-dimensional, conformal radiotherapy in patients with inoperable T1-3 N0 M0 non-small cell lung cancer.

Secondary

* Determine the toxicities of this regimen in these patients.
* Determine the rates of regional and distant disease recurrence in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the changes in pulmonary function after treatment in these patients.
* Assess the quality of life of patients after treatment.

OUTLINE: This is a multicenter, prospective study.

Patients undergo accelerated hypofractionated conformal radiotherapy 5 days a week for up to 3 weeks (15 doses) in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at week 3 of radiotherapy, at 1 month after completion of radiotherapy, and then every 4 months for 1 year.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage I or II peripheral disease

    * T1, N0, M0
    * T2 (≤ 5 cm), N0, M0
    * T3 (≤ 5 cm, chest wall primary tumor only), N0, M0
    * No T2-T3 primary tumors > 5 cm or any T1-T3 tumor of the mainstem bronchus involvement
    * No T1-T3 tumor in the lung apex (i.e., tumor in a position that will result in irradiation of the brachial plexus to the prescribed dose)
    * Hilar or mediastinal lymph nodes ≤ 1 cm considered N0
  * Any of the following primary cancer types:

    * Squamous cell carcinoma
    * Adenocarcinoma
    * Large cell carcinoma
    * Bronchioloalveolar cell carcinoma
    * Non-small cell carcinoma not otherwise specified
* Underlying physiological medical condition that prohibits surgery due to a low probability of tolerating general anesthesia, the operation, the postoperative recovery period, or the removal of adjacent functional lung (i.e., medically inoperable)
* Cytologic specimens obtained by brushing, washing, or needle aspiration of defined lesion allowed

  * If sputum cytology alone is used for diagnosis, it must be confirmed on a second specimen
* Must develop a radiotherapy plan that meets the dose-volume constraints for critical organs
* No ataxia telangiectasia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Able and willing to complete a quality of life questionnaire unless not literate in either English or French (i.e., a translator is required to comprehend the questions and reply)
* No active systemic, pulmonary, or pericardial infection
* No previous malignancy except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix.

  * Previous diagnosis of cancer that is free of recurrence and metastases for ≥ 2 years and, in the opinion of the treating physician, does not have a substantial risk of recurrence allowed (including prior lung cancer)

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the area of the primary tumor
* No prior or concurrent chemotherapy or immunotherapy for this tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-08-02 (Actual); Primary Completion 2012-02-28 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Local tumor control rate at 2 years | 2 years
  Overall tumor control rate will be assessed at 6 years

SECONDARY OUTCOMES:
Toxicity | 6 years
Disease recurrence rates | 6 years
Progression-free survival | 6 years
Overall survival | 6 years
Quality of life | 6 years
Changes in pulmonary function | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick CF Cheung, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Sergio L Faria, MD, PhD, Study Chair — Montreal General Hospital
Locations (19):
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheung P, Faria S, Ahmed S, Chabot P, Greenland J, Kurien E, Mohamed I, Wright JR, Hollenhorst H, de Metz C, Campbell H, Vu TT, Karvat A, Wai ES, Ung YC, Goss G, Shepherd FA, O'Brien P, Ding K, O'Callaghan C. Phase II study of accelerated hypofractionated three-dimensional conformal radiotherapy for stage T1-3 N0 M0 non-small cell lung cancer: NCIC CTG BR.25. J Natl Cancer Inst. 2014 Jul 29;106(8):dju164. doi: 10.1093/jnci/dju164. Print 2014 Aug. PMID 25074417